CLINICAL TRIAL: NCT05670483
Title: Use of Airway Pressure Release Ventilation in Morbidly Obese Patients Undergoing Open Heart Surgery to Improve Post Operative Pulmonary Outcomes
Brief Title: Use of Airway Pressure Release Ventilation in Morbidly Obese Patients Undergoing Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Alaaeldin Abdelmoneem Alhadidy, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU R 243/2022
Record Dates: First submitted 2022-12-08; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Pulmonary Atelectasis; Morbid Obesity; Pulmonary Complication
Keywords: APRV; Morbid Obesity; Cardiac surgery; Pulmonary Complications
MeSH Terms: conditions — Pulmonary Atelectasis; Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APRV group (Active Comparator): Group A: APRV group (30 Patients) Post operatively, Patients will be ventilated with APRV mode using GE Carescape R860 ventilator Initial Settings15
  1. P high at the P plateau (or desired P mean + 3cm H2O). keep P high below 30-35 cm H2O
  2. T high at 4-6 seconds
  3. P low at 0
  4. T low at 0.5 to 0.8 seconds.
  5. ATC (automatic tube compensation) on.
  6. FIO2: 40% Ventilator settings will be adjusted to keep Pco2 between 35-45 mmhg, PO2 > 60 mmhg on FIO2 < 50 % Once Patients are fully conscious and after complete recovery of reflexes with no postoperative bleeding nor hemodynamic instability, weaning of APRV will start as following, P-High will be lowered 2 or 3 cm of H2O pressure at a time, and T Low will be lengthened in 0.5-2.0 s increments, depending on patient tolerance. When the P-high reaches 10 cmH2O and the Thigh reaches 12-15 seconds, change the mode to pressure support (PS) mode PS of 7-8 cmH20 above PEEP of cmh2o then extubation.
  Interventions: Device: Use Of APRV mode of Ventilation
- Standard group (Active Comparator): Group B: Standard (control) group (30 Patients) Post-operatively, Patients will be ventilated with conventional Synchronized Intermittent Mandatory Ventilation (SIMV) volume control mode using GE Carescape R860 ventilator Initial Settings: 16
  1. Tidal Volume 6-8 ml/kg predicted body weight
  2. Respiratory rate (RR) 14 /min
  3. Positive end expiratory pressure (PEEP)= 5 cmH2o
  4. Pressure Support (PS) = 10 cmH2o
  5. Inspiratory time 1.4 Sec
  6. FIO2: 40% Ventilator settings will be adjusted to keep Pco2 between 35-45 mmhg, PO2 > 60 mmhg on FIO2 < 50 %
  Interventions: Device: Use of conventional Synchronized Intermittent Mandatory Ventilation (SIMV) volume control mode

INTERVENTIONS:
Device: Use Of APRV mode of Ventilation — Post operatively, Patients will be ventilated with APRV mode using GE Carescape R860 ventilator Initial Settings15
  1. P high at the P plateau (or desired P mean + 3cm H2O). keep P high below 30-35 cm H2O
  2. T high at 4-6 seconds
  3. P low at 0
  4. T low at 0.5 to 0.8 seconds.
  5. ATC (automatic tube compensation) on.
  6. FIO2: 40% Ventilator settings will be adjusted to keep Pco2 between 35-45 mmhg, PO2 > 60 mmhg on FIO2 < 50 % Once Patients are fully conscious and after complete recovery of reflexes with no postoperative bleeding nor hemodynamic instability, weaning of APRV will start as following, P-High will be lowered 2 or 3 cm of H2O pressure at a time, and T Low will be lengthened in 0.5-2.0 s increments, depending on patient tolerance. When the P-high reaches 10 cmH2O and the Thigh reaches 12-15 seconds, change the mode to pressure support (PS) mode PS of 7-8 cmH20 above PEEP of cmh2o then extubation.
  Arms: APRV group
Device: Use of conventional Synchronized Intermittent Mandatory Ventilation (SIMV) volume control mode — Post-operatively, Patients will be ventilated with conventional Synchronized Intermittent Mandatory Ventilation (SIMV) volume control mode using GE Carescape R860 ventilator Initial Settings: 16
  1. Tidal Volume 6-8 ml/kg predicted body weight
  2. Respiratory rate (RR) 14 /min
  3. Positive end expiratory pressure (PEEP)= 5 cmH2o
  4. Pressure Support (PS) = 10 cmH2o
  5. Inspiratory time 1.4 Sec
  6. FIO2: 40% Ventilator settings will be adjusted to keep Pco2 between 35-45 mmhg, PO2 > 60 mmhg on FIO2 < 50 % Once Patients are fully conscious and after complete recovery of reflexes with no postoperative bleeding nor hemodynamic instability, weaning of mechanical ventilation will be done by switching the ventilation to pressure support (PS) mode PS of 7-8 cmH20 above PEEP of cmh2o then extubation.
  Arms: Standard group

SUMMARY:
The goal of this Randomized Clinical trial is to to investigate if the use of Air Pressure Release Ventilation in morbidly obese patients undergoing open heart surgery will improve post operative pulmonary outcomes 60 Patients will be randomized into two groups according to the mode of ventilation used into: Group A: airway pressure release ventilation (APRV) group (30 Patients) Group B: Standard (control) group (30 Patients) Post-operatively, Patients will be ventilated with conventional Synchronized Intermittent Mandatory Ventilation (SIMV) volume control mode

DETAILED DESCRIPTION:
Obesity is an ongoing worldwide problem, and as such, weight-related issues arise especially in the intensive care unit (ICU). Morbid obesity adversely affects physiology; restricted thoracic movement and increased intra-abdominal pressure leads to reduced lung volumes and compliance resulting frequently in atelectasis, ventilation-perfusion mismatch.

Cardiac surgical patients are at particular risk for PPCs. The use of cardiopulmonary bypass (CPB) is responsible for a systemic inflammatory response and oxidative stress, leading to pulmonary ischemia-reperfusion injury. Mechanical ventilation frequently is disrupted during CPB, thus inducing atelectasis. Some proposed mechanisms are leukocyte activation, fluid accumulation in the lung and atelectasis.

Atelectasis is a highly prevalent pulmonary complication in patients undergoing cardiac surgery with cardiopulmonary bypass (CPB) and an important cause of postoperative hypoxemia. Pulmonary collapse occurs early after the induction of anesthesia and persists for several days postoperatively. Studies based on thoracic computed tomography (CT) have shown that pulmonary collapse is mainly distributed to the dependent regions close to the diaphragm and may encompass up to 35% of the overall lung parenchyma which predispose to pneumonia.

This impairment of lung function, particularly oxygenation of the blood, is a common and potentially serious complication after cardiac surgery. It has been shown to persist for as long as one week after the operation.

In obese patients, the functional residual capacity (FRC) and lung compliance are reduced, and thus the elastic work of breathing (WOB) is elevated. By applying continuous positive airway pressure (CPAP), the FRC is restored, and inspiration starts from a more favorable pressure-volume relationship, facilitating spontaneous ventilation, and improves oxygenation.

APRV was originally described as a mode to treat acute lung injury in patients and attempt to maintain the level of airway pressure without reducing cardiac function, delivering mechanical breaths without excessive airway pressure and allowing unrestricted spontaneous ventilation. 6 APRV is essentially a high-level continuous positive airway pressure (CPAP) mode that is terminated for a very brief period of time. It is this short release period that allows carbon dioxide to be cleared. The lengthy time during which the high-level CPAP is present results in substantial recruitment of alveoli of markedly different regional time constants, at rather low gas flow rates and lower airway pressures. The establishment of intrinsic PEEP by the short release time enhances oxygenation. Carbon dioxide clearance is aided by recruitment of the patient's lung at close to total lung capacity; elastic recoil creates large volume gas flow during the release period.

Recent advances in the understanding of the respiratory physiologic alterations in the obese patient suggest that ''open lung'' ventilation approaches such as APRV recruit lung alveolar volumes without exacerbating lung injury and maintain acceptable gas exchange. Given the spontaneous nature of the mode, it is hypothesized that there should be no need for continuous infusions of neuromuscular blocking agents in patients placed on this mode of ventilation.

This may result in a shorter duration of intensive care unit (ICU) stay. Furthermore, because patients may be ventilated at lower airway pressures than are required with cyclic ventilation, there may be a reduced need for pressor support of hemodynamics to ensure oxygen delivery which is favorable in cardiac surgical patients.

So, the investigators hypothesize that APRV may be a preferred mode of ventilation in morbidly obese patients after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 y.
* Scheduled for open heart Surgery with cardiopulmonary bypass (CPB) pump.
* Class III Obesity (Morbid obesity): BMI ≥ 40.0 kg/m².

Exclusion Criteria:

* Patients with obstructive lung disease (asthma or chronic obstructive pulmonary disease).
* Pneumothorax or Surgical emphysema.
* Mechanical ventilation prior to the operation.
* Patient Refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-03 (Actual); Primary Completion 2023-05-03 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
PO2/FIO2 (P/F) ratio | up to 3 days
  Will be recorded at admission, 6 hours,12 hours, 24 hours and 48 hours
Time of mechanical ventilation | up to 3 days
  Hours of Mechanical ventilation

SECONDARY OUTCOMES:
Need for Non-Invasive ventilation (NIV) | up to 3 days
  Need of high flow nasal cannula (HFNC) or Non-Invasive continuous positive airway pressure (NICPAP)
Occurrence Respiratory complications | up to 1 week
  Occurrence of Pneumonia identified by clinical signs, chest Xray and lung ultrasound
Effect on Blood pressure | up to 1 day
  Mean arterial systemic blood pressure (MAP) recorded at admission, 6 hours, 12 hours and 24 hours
Need for Vasopressors and Inotropes | up to 1 day
  Vasopressors and Inotropes needs guided by Vasoactive-Inotrope score (VIS) measured at admission, 6 hours, 12 hours and 24 hours
length of ICU stay | up to 3 days
  Duration of patient stays in ICU in days
length of Hospital stay | up to 10 days
  Duration of hospital stay after surgery in days.
Mortality | up to 30 days
  Post operative Death

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiothoracic Academy, Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Villavicencio MA, Sundt TM 3rd, Daly RC, Dearani JA, McGregor CG, Mullany CJ, Orszulak TA, Puga FJ, Schaff HV. Cardiac surgery in patients with body mass index of 50 or greater. Ann Thorac Surg. 2007 Apr;83(4):1403-11. doi: 10.1016/j.athoracsur.2006.10.076. PMID 17383347
- [Background] Ranucci M, Ballotta A, La Rovere MT, Castelvecchio S; Surgical and Clinical Outcome Research (SCORE) Group. Postoperative hypoxia and length of intensive care unit stay after cardiac surgery: the underweight paradox? PLoS One. 2014 Apr 7;9(4):e93992. doi: 10.1371/journal.pone.0093992. eCollection 2014. PMID 24709952
- [Background] Neves FH, Carmona MJ, Auler JO Jr, Rodrigues RR, Rouby JJ, Malbouisson LM. Cardiac compression of lung lower lobes after coronary artery bypass graft with cardiopulmonary bypass. PLoS One. 2013 Nov 11;8(11):e78643. doi: 10.1371/journal.pone.0078643. eCollection 2013. PMID 24244331
- [Background] Daoud EG. Airway pressure release ventilation. Ann Thorac Med. 2007 Oct;2(4):176-9. doi: 10.4103/1817-1737.36556. PMID 19727373
- [Background] Ge H, Lin L, Xu Y, Xu P, Duan K, Pan Q, Ying K. Airway Pressure Release Ventilation Mode Improves Circulatory and Respiratory Function in Patients After Cardiopulmonary Bypass, a Randomized Trial. Front Physiol. 2021 Jun 3;12:684927. doi: 10.3389/fphys.2021.684927. eCollection 2021. PMID 34149459
- [Background] Testerman GM, Breitman I, Hensley S. Airway pressure release ventilation in morbidly obese surgical patients with acute lung injury and acute respiratory distress syndrome. Am Surg. 2013 Mar;79(3):242-6. PMID 23461947
- [Background] Kaplan LJ, Bailey H, Formosa V. Airway pressure release ventilation increases cardiac performance in patients with acute lung injury/adult respiratory distress syndrome. Crit Care. 2001 Aug;5(4):221-6. doi: 10.1186/cc1027. Epub 2001 Jul 2. PMID 11511336
- [Background] Bonatti G, Robba C, Ball L, Silva PL, Rocco PRM, Pelosi P. Controversies when using mechanical ventilation in obese patients with and without acute distress respiratory syndrome. Expert Rev Respir Med. 2019 May;13(5):471-479. doi: 10.1080/17476348.2019.1599285. Epub 2019 Apr 5. PMID 30919705
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Manjunath V, Reddy BG, Prasad SR. Is airway pressure release ventilation, a better primary mode of post-operative ventilation for adult patients undergoing open heart surgery? A prospective randomised study. Ann Card Anaesth. 2021 Jul-Sep;24(3):288-293. doi: 10.4103/aca.ACA_98_20. PMID 34269256
- [Background] Sawano Y, Miyazaki M, Shimada H, Kadoi Y. Optimal fentanyl dosage for attenuating systemic hemodynamic changes, hormone release and cardiac output changes during the induction of anesthesia in patients with and without hypertension: a prospective, randomized, double-blinded study. J Anesth. 2013 Aug;27(4):505-11. doi: 10.1007/s00540-012-1552-x. Epub 2013 Jan 12. PMID 23314694
- [Background] Members of the Working Party; Nightingale CE, Margarson MP, Shearer E, Redman JW, Lucas DN, Cousins JM, Fox WT, Kennedy NJ, Venn PJ, Skues M, Gabbott D, Misra U, Pandit JJ, Popat MT, Griffiths R; Association of Anaesthetists of Great Britain; Ireland Society for Obesity and Bariatric Anaesthesia. Peri-operative management of the obese surgical patient 2015: Association of Anaesthetists of Great Britain and Ireland Society for Obesity and Bariatric Anaesthesia. Anaesthesia. 2015 Jul;70(7):859-76. doi: 10.1111/anae.13101. Epub 2015 May 7. PMID 25950621
- [Background] Alwardt CM, Redford D, Larson DF. General anesthesia in cardiac surgery: a review of drugs and practices. J Extra Corpor Technol. 2005 Jun;37(2):227-35. PMID 16117465
- [Background] Modrykamien A, Chatburn RL, Ashton RW. Airway pressure release ventilation: an alternative mode of mechanical ventilation in acute respiratory distress syndrome. Cleve Clin J Med. 2011 Feb;78(2):101-10. doi: 10.3949/ccjm.78a.10032. PMID 21285342
- [Result] Fischer MO, Brotons F, Briant AR, Suehiro K, Gozdzik W, Sponholz C, Kirkeby-Garstad I, Joosten A, Nigro Neto C, Kunstyr J, Parienti JJ, Abou-Arab O, Ouattara A; VENICE study group. Postoperative Pulmonary Complications After Cardiac Surgery: The VENICE International Cohort Study. J Cardiothorac Vasc Anesth. 2022 Aug;36(8 Pt A):2344-2351. doi: 10.1053/j.jvca.2021.12.024. Epub 2021 Dec 25. PMID 35094928